CLINICAL TRIAL: NCT02683122
Title: Improvement of Diagnosis of Hospital Acquired Pneumonia (HAP) Based on Early Organ Dysfunction
Brief Title: The DIPOD Study (Diagnosis Improvement of Pneumonia by Organ Dysfunction)
Acronym: DIPOD
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: P15-37816003/2015-NI
Record Dates: First submitted 2016-01-11; First posted 2016-02-17 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Organ dysfunction scores; Pneumonia, Ventilator-Associated; Intensive care units
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The place of analysis of organ dysfunction in relation to the diagnosis of nosocomial pneumonia in intensive care is not yet defined.

DETAILED DESCRIPTION:
New onset of pulmonary infiltrates, fever, and an increase in white blood cell (WBC) count accompanied by purulent tracheal secretions are clinically indicative of hospital-associated pneumonia (HAP). The low specificity and sensibility of diagnostic tests for HAP, however, tends to result in an extremely high incidence of missed diagnoses and may lay to high mortality.

The place of analysis of organ dysfunction in relation to the diagnosis of nosocomial pneumonia in intensive care is not yet defined, because early organ dysfunction may be the first symptoms noted by clinicians.

ELIGIBILITY:
Inclusion Criteria:

Patients after cardiac/thoracic surgery with suspicion of HAP defined by the presence of the following criteria:

* new onset of pulmonary infiltrates,
* fever >38,3°C,
* increase in white blood cell (WBC) count
* purulent tracheal secretions
* but also:
* increased use of catecholamine,
* need of volemic expansion,
* depletion inability,
* confusion,
* hepatic perturbation with increased gamma-glutamyl transpeptidase (GGT)>2N or alkaline phosphatase (ALP) >1.5 N, or bilirubin >1.5N, or aminotransferase (AST or ALT>2 N).

Exclusion Criteria:

* child,
* pregnancy,
* end of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Intensive care unit after cardiac and/or thoracic surgery with a clinical suspicion of HAP
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Area under the ROC curve of the CPIS score | the previous 12 hours up to performance of pulmonary bacteriological samples
  The CPIS score is based on six variables:
  * Fever
  * Leukocytosis
  * Tracheal aspirates
  * Oxygenation
  * Radiographic infiltrates
  * Cult of tracheal aspirates

SECONDARY OUTCOMES:
Area under the ROC curve of increased use of catecholamine and their positive and negative predictive values | the previous 12 hours up to performance of pulmonary bacteriological samples
  Sensibility (%) and specificity (%) increased use of catecholamine
Area under the ROC curve of increased need a volemic expansion and their positive and negative predictive values | the previous 12 hours up to performance of pulmonary bacteriological samples
  Sensibility (%) and specificity (%) increased need a volemic expansion
Area under the ROC curve of depletion inability and their positive and negative predictive values | the previous 12 hours up to performance of pulmonary bacteriological samples
  Sensibility (%) and specificity (%) of depletion inability
Area under the ROC curve of confusion and their positive and negative predictive values | the previous 12 hours up to performance of pulmonary bacteriological samples
  Sensibility (%) and specificity (%) of confusion
Area under the ROC curve of hepatic perturbation and their positive and negative predictive values | the previous 12 hours up to performance of pulmonary bacteriological samples
  Sensibility (%) and specificity (%) of hepatic perturbation defined by increased gamma-glutamyl transpeptidase (CGT) and or alkaline phosphatase >1,5 N and or bilirubin >1,5 N or aminotransferase (AST or ALT >2 N)
Mortality | 28 days
  Mortality during ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: TALNA KORTCHINSKY, MD, Principal Investigator — Centre Chirurgical Marie Lannelongue
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500
- [Background] Calandra T, Cohen J; International Sepsis Forum Definition of Infection in the ICU Consensus Conference. The international sepsis forum consensus conference on definitions of infection in the intensive care unit. Crit Care Med. 2005 Jul;33(7):1538-48. doi: 10.1097/01.ccm.0000168253.91200.83. PMID 16003060